CLINICAL TRIAL: NCT04111224
Title: Evaluation of Pentraxin3 as an Early Marker in the Diagnosis of Ventilator-associated Pneumonia
Brief Title: Evaluation of pentraxin3 as a Marker for Ventilator Associated Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham mohamed ahmed abdelsater, resident dr, Assiut University
Other Study IDs: PTX 3 as a marker for VAP
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pentraxin 3 marker — Assess the role of pentraxin3 (PTX3) in the early diagnosis of ventilator-associated pneumonia (VAP).

SUMMARY:
This study will assess the role of pentraxin3 (PTX3) in the early diagnosis of ventilator-associated pneumonia (VAP) and the detection of antibiotic sensitivity for different organisms isolated from tracheal aspirate.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is a type of hospital-acquired pneumonia that occurs more than 48h after endotracheal intubation. This can be further classified into early onset (within the first 96 hours of mechanical ventilation (MV) and late onset (more than 96 hours after the initiation of MV), which is more commonly attributable to multidrug-resistant pathogens Ventilator associated pneumonia is common in critical care patients and is responsible for around half of all antibiotics given to patients in intensive care units. International Nosocomial Infection Control Consortium suggest that the overall rate of VAP is 13.6 per 1000 ventilator days. However, the individual rate varies according to patient group, risk factors and hospital setting. The average time taken to develop VAP from the initiation of MV is around 5 to 7 days, with a mortality rate quoted as between 24% and 76%.

The key to the development of VAP is the presence of an endotracheal tube (EET) or tracheostomy, both of which interfere with the normal anatomy and physiology of respiratory tract, specifically the functional mechanisms involved in clearing secretion (cough and mucociliary action).

Intubated patients have a reduced level of consciousness that impairs voluntary clearance of secretions, which may then pool in the oropharynx. This leads to the macro aspiration and micro aspiration of contaminated oropharyngeal secretions that are rich in harmful pathogens. Normal oral flora starts to proliferate and are able to pass along the tracheal tube, forming an antibiotic-resistant biofilm which eventually reaches the lower airways.

Critically unwell patients exhibit an impaired ability to mount an immune response to these pathogens, leading to the development of a pneumonia.

Early-onset VAP, occurring within the first four days of MV, is usually caused by antibiotic-sensitive community-acquired bacteria such as Hemophilus and Streptococcus. VAP developing more than 5 days after initiation of MV is usually caused by multidrug-resistant bacteria such as Pseudomonas aeruginosa.

The clinical pulmonary infection score (CPIS) based on variables (fever, leukocytosis, tracheal aspirates, oxygenation radiographic infiltrates). CPIS is helpful to diagnosis VAP in patient but it is not sufficient for definite diagnosis.

The accurate diagnosis of VAP in children and adults is still an unsolved problem, delayed diagnosis of VAP and subsequent delay in initiating appropriate therapy may cause worse outcomes in patients with VAP. On the other hand, an incorrect diagnosis may lead to unnecessary treatment and subsequent complications that are related to therapy. Over-treatment with antibiotics increases clinical risks such as Clostridium difficile-associated colitis and antibiotic resistance.

Several criteria have been proposed for diagnosing VAP in clinical settings, including clinical manifestations, imaging techniques, methods to obtain and interpret bronchoalveolar specimens, and biomarkers of host response. However, there is no acceptable gold standard modality yet and the accuracy of these methods in diagnosing VAP is controversial.

Microbiological analysis and identification of organisms may take 48-72 h, false-negative results may occur as a result of concomitant or previous antibiotic treatment, whereas false positives may represent colonization or sampling errors. Biomarkers have been seen as a potential avenue for improving speed and accuracy of clinical diagnosis, or to allow withdrawal of therapy because of the clinical resolution of VAP.

Pentraxins are phylogenetically conserved proteins characterized by a multimeric structure and divided into short (C -reactive protein (CRP) and serum amyloid P component) and long pentraxins.

PTX3 is the first identified member of the long pentraxin subfamily. It can be rapidly produced and released by mononuclear phagocytes, neutrophils, epithelial and endothelial cells in response to primary inflammatory signals (IL-1, and TNF-α).

Pentraxin3 (PTX3) is an acute-phase inflammatory mediator whose levels increase rapidly in inflammatory and infectious conditions. Increased PTX3 levels are correlated with the severity of lung injury and infection.

ELIGIBILITY:
Inclusion Criteria:

* study will be conducted on adult patients >18 years who will have VAP in intensive care unit (ICU) of chest department of Assiut university hospital.

Exclusion Criteria:

* Patients with age <18 years .
* Patients with any hospital acquired infections other than VAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients will be included in the study, the first sample will be taken in the first day of the endotracheal intubation as a control sample then the second sample will be the part the first sample patients who will develop VAP (>48 h of endotracheal intubation).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Assess the role of pentraxin3 (PTX3) in the early diagnosis of ventilator-associated pneumonia (VAP). | Baseline
  Pentraxin3 (PTX3) is an acute-phase inflammatory mediator whose levels increase rapidly in inflammatory and infectious conditions. Increased PTX3 levels are correlated with the severity of lung injury and infection.

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Abdelsater, resident dr, Principal Investigator — Assiut University; Monazzma A Fadel, professor, Study Director — Assiut University; Amal M Hosni, lecturer, Study Director — Assiut University